CLINICAL TRIAL: NCT06317012
Title: Assessment Of Computer-Aided Design/Manufacturing for Le Fort I Osteotomy and 3D-customized Titanium Plate in Orthognathic Surgery (Clinical Trial)
Brief Title: Computer-Aided Design/Manufacturing for Le Fort I Osteotomy and 3D-customized Titanium Plate in Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0407-03/2022
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Le Fort; I

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Le Fort I osteotomy (Experimental)
  Interventions: Procedure: Le Fort I osteotomy using CAD CAM surgical guide and 3Dcustomized plate

INTERVENTIONS:
Procedure: Le Fort I osteotomy using CAD CAM surgical guide and 3Dcustomized plate — Le Fort I osteotomy will be performed with the aid of a surgical guide through the mucosal incision at the maxillary vestibule region, providing adequate surgical exposure.
  The planned position will be obtained using a customized titanium plate for precise maxillary position and fixation as planned virtually on the software.

SUMMARY:
Background: In orthognathic surgery, virtual planning is gradually taking over in clinical practice. To start with, virtual surgery planning (VSP) is believed to be less time-consuming and less expensive than conventional surgery planning (CSP). Moreover, the improved visualization of craniofacial deformities, such as occlusal canting and asymmetries, is a further advantage. Aim: To assess the result of Le Fort I osteotomy using CAD/CAM and 3Dcustomized titanium plate with virtual planning in orthognathic surgery. Materials and Methods: 8 patients with vertical maxillary excess will be included in the study. Le Fort I osteotomy using CAD CAM surgical guide and 3Dcustomized plate will be done for the study group. All patients will be followed clinically and radiographically for one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-syndromic dentofacial deformity requiring isolated Le Fort I with or without bimaxillary osteotomy.
* Patients with good oral hygiene.
* Class II or III malocclusion.
* Patients who were scheduled to undergo a CT scan as a part of their diagnosis and treatment

Exclusion Criteria:

* Patients with acute infection at the surgery site.
* Patient with Systemic disorders contraindicating surgery.
* Smokers.
* Alcohol or drug abuse is prohibited.
* patients who suffered from craniofacial syndrome;
* patients who had previous orthognathic surgery;
* patients who had previous maxillary or mandibular trauma

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain | 2nd and 7th days
  pain will be scored using visual analogue scale. it ranges from 0 to 10, 0 mean no pain and 10 means severe pain
change in edema | 2nd and 7th days
  it was evaluated by its ability to pit. The examiner's fingers will press into the dependent area for 5 seconds, and the pitting will be graded on a scale of +1 to+4.
Change in post operative osteotomy position | Immediate post operative
  Computed tomography (CT) will be used immediately postoperative to assess surgical position by comparing the clinical results with the virtually planned outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt